CLINICAL TRIAL: NCT04964843
Title: A Pilot Study of N-acetylcysteine for Alcohol Use Disorder
Brief Title: A Study of NAC for AUD
Acronym: NAC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Null results were posted from a neurometabolite study and a recent trial for AUD. Study may resume if more positive data emerge.
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0000
Record Dates: First submitted 2021-06-17; First posted 2021-07-16 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Arm 1: n-acetylcysteine. 25 participants randomly selected Arm 2: placebo. 25 participants randomly selected
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- N-acetylcysteine (Experimental): 25 participants randomly selected to receive 1500 milligrams of oral n-acetylcysteine twice daily for 7 weeks.
  Interventions: Drug: N-acetylcysteine
- Placebo (Placebo Comparator): 25 participants randomly selected to receive placebo twice daily for 7 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine is an FDA approved medication that is used to treat acetaminophen overdose.
  Arms: N-acetylcysteine
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This proposed pilot study aims to assess the effects of N-acetylcysteine (NAC) on alcohol use disorder (AUD). Despite promising preliminary research, no investigations to date have focused on NAC with alcohol use as the primary aim or on individuals specifically seeking treatment for AUD. The present proposal is an 7-week randomized, double-blind, placebo-controlled study of 3000mg of NAC in up to 50 participants (25 NAC, 25 placebo).

The primary aim of the current study is to establish feasibility, dropout rate, and estimate the standard deviation of the outcome measures in order to estimate the required sample for a fully powered clinical trial and to refine the final measures for use in the fully powered clinical trial. Additionally, this study will explore preliminary efficacy signal of NAC.

DETAILED DESCRIPTION:
Alcohol abuse is responsible for 1 in 10 deaths among working age adults in the U.S. and costs ~$249 billion annually. Currently approved medications for alcohol use disorder (AUD) exert only small to medium effects on drinking, with estimates indicating 12 to 20 drinkers need to be treated for one of them to benefit from the two leading medications, acamprosate and naltrexone. Thus, many patients do not benefit from current pharmacotherapies for AUD.

N-acetylcysteine (NAC) is one promising pharmacotherapy that is well-tolerated, safe, and exhibits preliminary evidence across a number of psychiatric and neurological disorders. NAC is available over the counter, has been used all over the world for a variety of conditions, most notably for its 1985 FDA approved use as an antidote for acetaminophen overdose.

The NAC dosage was selected as most prior studies in addiction have used 2400-3000mg and even studies up to 3600mg have found it was well-tolerated. Many studies using doses in this range achieved clinically significant improvements, including a study of NAC for smoking cessation which used 3000mg. 7 weeks was selected rather than 12 weeks or longer duration because this within the range of prior clinical trials of NAC (most are 8-12 weeks) and is fitting for the goals of this pilot trial seeking to establish feasibility and sample size for a larger clinical trial. It is beyond the primary aims of this study and the resources of the team to seek longer term outcomes (e.g., drinking at 6 months; https://www.fda.gov/media/91222/download).

ELIGIBILITY:
Inclusion criteria:

1. Greater than or equal to 18 years of age
2. Meets DSM-V criteria for alcohol use disorder on the SCID-5
3. MHS Healthcare Beneficiary

NOTE. While we are recruiting explicitly from the Addiction Treatment Services (ATS) patient population, we do not require that they are currently receiving treatment at ATS. For participants that are not currently in care we will provide them with resources to pursue psychotherapy while engaged in our study as outlined in the interview treatment questions and physical and mental health resource document.

Exclusion criteria:

1. Lifetime clinical diagnosis of schizophrenia or bipolar disorder
2. Currently receiving medication for the treatment of alcohol use disorder including oral or injectable naltrexone (ReVia, Vivitrol), disulfiram (Antabuse), and acamprosate (Campral).
3. Pregnancy
4. Lack of English fluency sufficient to complete study measures.
5. Trying to get pregnant in the next 4 months.
6. Hospitalized because of alcohol use in the past 12 months.
7. History of seizures or delirium tremens.
8. History of liver disease
9. Diagnosis of a neurocognitive disorder (e.g., dementia, alzheimer's, mental retardation).
10. Individuals who were never enrolled into Addiction Treatment Services

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Change in total drinking days | 7 weeks
  Change in total drinking days will be assessed with the Timeline Follow Back alcohol use assessment
Change in drinks per drinking day | 7 weeks
  Change in drinks per drinking day will be assessed with the Timeline Follow Back alcohol use assessment

SECONDARY OUTCOMES:
Change in alcohol cue-reactivity | 7 weeks
  Change in alcohol cue-reactivity will be assessed with a task in which participants are exposed to stimuli associated with alcohol
Change in alcohol demand | 7 weeks
  Change in alcohol demand will be assessed with the alcohol purchase task
Change in alcohol craving | 7 weeks
  Change in alcohol craving will be assessed with the Penn Alcohol Craving Scale, a 5-item measure of craving for alcohol over the past week. Scores range from 0 to 30, higher scores indicate more alcohol craving.

OTHER OUTCOMES:
Change in response inhibition | 7 weeks
  Change in response inhibition will be assessed with the Stop Signal Task.
Change in working memory | 7 weeks
  Change in working memory will be assessed with the N-back task (2 back and 3 back)
Change in executive functioning | 7 weeks
  Change in executive functioning will be assessed with the Trail Making Task
Change in depression symptoms | 7 weeks
  Change in depression symptoms will be assessed with the Montgomery-Åsberg Depression Rating Scale (MADRS), a 10-item questionnaire assessing depression symptoms. Scores range from 0-60, higher scores indicate more depression symptoms
Change in anxiety symptoms | 7 weeks
  Change in anxiety symptoms will be assessed with the Generalized Anxiety Disorder Screener (GAD-7), a 7-item self-report measure assessing symptoms of generalized anxiety. Scores range from 0-21, higher scores indicate more anxiety symptoms.
Change in anxiety symptoms | 7 weeks
  Change in anxiety symptoms will be assessed with the Social Interaction Anxiety Scale (SIAS-6), a 6-item measure of social interaction anxiety. Scores range from 0-24 where higher scores indicate higher anxiety.
Change in anxiety symptoms | 7 weeks
  Change in anxiety symptoms will be assessed with the Social Phobia Scale (SPS-6), a 6-item measure of social phobia anxiety. Scores range from 0-24 where higher scores indicate higher anxiety.
Change in total marijuana use days | 7 weeks
  Change in total marijuana use days will be assessed with the Timeline Follow Back marijuana use assessment in the subset of individuals who use marijuana.
Change in total cigarette use days | 7 weeks
  Change in total cigarette use days will be assessed with the Timeline Follow Back cigarette use assessment in the subset of individuals who use cigarettes.
Change in cigarettes per day | 7 weeks
  Change in cigarettes per day will be assessed with the Timeline Follow Back cigarette use assessment in the subset of individuals who use cigarettes.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stahre M, Roeber J, Kanny D, Brewer RD, Zhang X. Contribution of excessive alcohol consumption to deaths and years of potential life lost in the United States. Prev Chronic Dis. 2014 Jun 26;11:E109. doi: 10.5888/pcd11.130293. PMID 24967831
- [Background] Jonas DE, Amick HR, Feltner C, Bobashev G, Thomas K, Wines R, Kim MM, Shanahan E, Gass CE, Rowe CJ, Garbutt JC. Pharmacotherapy for adults with alcohol use disorders in outpatient settings: a systematic review and meta-analysis. JAMA. 2014 May 14;311(18):1889-900. doi: 10.1001/jama.2014.3628. PMID 24825644
- [Background] Minarini A, Ferrari S, Galletti M, Giambalvo N, Perrone D, Rioli G, Galeazzi GM. N-acetylcysteine in the treatment of psychiatric disorders: current status and future prospects. Expert Opin Drug Metab Toxicol. 2017 Mar;13(3):279-292. doi: 10.1080/17425255.2017.1251580. Epub 2016 Nov 2. PMID 27766914
- [Background] Fernandes BS, Dean OM, Dodd S, Malhi GS, Berk M. N-Acetylcysteine in depressive symptoms and functionality: a systematic review and meta-analysis. J Clin Psychiatry. 2016 Apr;77(4):e457-66. doi: 10.4088/JCP.15r09984. PMID 27137430
- [Background] Burnett EJ, Chandler LJ, Trantham-Davidson H. Glutamatergic plasticity and alcohol dependence-induced alterations in reward, affect and cognition. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Feb 4;65:309-20. doi: 10.1016/j.pnpbp.2015.08.012. Epub 2015 Sep 1. PMID 26341050
- [Background] Dean O, Giorlando F, Berk M. N-acetylcysteine in psychiatry: current therapeutic evidence and potential mechanisms of action. J Psychiatry Neurosci. 2011 Mar;36(2):78-86. doi: 10.1503/jpn.100057. PMID 21118657
- [Background] Legastelois R, Botia B, Coune F, Jeanblanc J, Naassila M. Deciphering the relationship between vulnerability to ethanol-induced behavioral sensitization and ethanol consumption in outbred mice. Addict Biol. 2014 Mar;19(2):210-24. doi: 10.1111/adb.12104. Epub 2013 Oct 29. PMID 24164956
- [Background] Morais-Silva G, Alves GC, Marin MT. N-acetylcysteine treatment blocks the development of ethanol-induced behavioural sensitization and related DeltaFosB alterations. Neuropharmacology. 2016 Nov;110(Pt A):135-142. doi: 10.1016/j.neuropharm.2016.07.009. Epub 2016 Jul 9. PMID 27401790
- [Background] Reyes RC, Cittolin-Santos GF, Kim JE, Won SJ, Brennan-Minnella AM, Katz M, Glass GA, Swanson RA. Neuronal Glutathione Content and Antioxidant Capacity can be Normalized In Situ by N-acetyl Cysteine Concentrations Attained in Human Cerebrospinal Fluid. Neurotherapeutics. 2016 Jan;13(1):217-25. doi: 10.1007/s13311-015-0404-4. PMID 26572666
- [Background] Lebourgeois S, Gonzalez-Marin MC, Jeanblanc J, Naassila M, Vilpoux C. Effect of N-acetylcysteine on motivation, seeking and relapse to ethanol self-administration. Addict Biol. 2018 Mar;23(2):643-652. doi: 10.1111/adb.12521. Epub 2017 May 30. PMID 28557352
- [Background] Schneider R Jr, Santos CF, Clarimundo V, Dalmaz C, Elisabetsky E, Gomez R. N-acetylcysteine prevents behavioral and biochemical changes induced by alcohol cessation in rats. Alcohol. 2015 May;49(3):259-63. doi: 10.1016/j.alcohol.2015.01.009. Epub 2015 Feb 13. PMID 25771148
- [Background] Quintanilla ME, Rivera-Meza M, Berrios-Carcamo P, Salinas-Luypaert C, Herrera-Marschitz M, Israel Y. Beyond the "First Hit": Marked Inhibition by N-Acetyl Cysteine of Chronic Ethanol Intake But Not of Early Ethanol Intake. Parallel Effects on Ethanol-Induced Saccharin Motivation. Alcohol Clin Exp Res. 2016 May;40(5):1044-51. doi: 10.1111/acer.13031. Epub 2016 Apr 8. PMID 27062046
- [Background] Schneider R Jr, Bandiera S, Souza DG, Bellaver B, Caletti G, Quincozes-Santos A, Elisabetsky E, Gomez R. N-acetylcysteine Prevents Alcohol Related Neuroinflammation in Rats. Neurochem Res. 2017 Aug;42(8):2135-2141. doi: 10.1007/s11064-017-2218-8. Epub 2017 Mar 16. PMID 28303497
- [Background] Morley KC, Baillie A, Van Den Brink W, Chitty KE, Brady K, Back SE, Seth D, Sutherland G, Leggio L, Haber PS. N-acetyl cysteine in the treatment of alcohol use disorder in patients with liver disease: Rationale for further research. Expert Opin Investig Drugs. 2018 Aug;27(8):667-675. doi: 10.1080/13543784.2018.1501471. Epub 2018 Aug 1. PMID 30019966
- [Background] Squeglia LM, Baker NL, McClure EA, Tomko RL, Adisetiyo V, Gray KM. Alcohol use during a trial of N-acetylcysteine for adolescent marijuana cessation. Addict Behav. 2016 Dec;63:172-7. doi: 10.1016/j.addbeh.2016.08.001. Epub 2016 Aug 4. PMID 27521979
- [Background] Squeglia LM, Tomko RL, Baker NL, McClure EA, Book GA, Gray KM. The effect of N-acetylcysteine on alcohol use during a cannabis cessation trial. Drug Alcohol Depend. 2018 Apr 1;185:17-22. doi: 10.1016/j.drugalcdep.2017.12.005. Epub 2018 Feb 1. PMID 29413434
- [Background] Gray KM, Carpenter MJ, Baker NL, DeSantis SM, Kryway E, Hartwell KJ, McRae-Clark AL, Brady KT. A double-blind randomized controlled trial of N-acetylcysteine in cannabis-dependent adolescents. Am J Psychiatry. 2012 Aug;169(8):805-12. doi: 10.1176/appi.ajp.2012.12010055. PMID 22706327
- [Background] Gray KM, Sonne SC, McClure EA, Ghitza UE, Matthews AG, McRae-Clark AL, Carroll KM, Potter JS, Wiest K, Mooney LJ, Hasson A, Walsh SL, Lofwall MR, Babalonis S, Lindblad RW, Sparenborg S, Wahle A, King JS, Baker NL, Tomko RL, Haynes LF, Vandrey RG, Levin FR. A randomized placebo-controlled trial of N-acetylcysteine for cannabis use disorder in adults. Drug Alcohol Depend. 2017 Aug 1;177:249-257. doi: 10.1016/j.drugalcdep.2017.04.020. Epub 2017 Jun 10. PMID 28623823
- [Background] LaRowe SD, Kalivas PW, Nicholas JS, Randall PK, Mardikian PN, Malcolm RJ. A double-blind placebo-controlled trial of N-acetylcysteine in the treatment of cocaine dependence. Am J Addict. 2013 Sep-Oct;22(5):443-52. doi: 10.1111/j.1521-0391.2013.12034.x. Epub 2013 May 15. PMID 23952889
- [Background] Costa DLC, Diniz JB, Requena G, Joaquim MA, Pittenger C, Bloch MH, Miguel EC, Shavitt RG. Randomized, Double-Blind, Placebo-Controlled Trial of N-Acetylcysteine Augmentation for Treatment-Resistant Obsessive-Compulsive Disorder. J Clin Psychiatry. 2017 Jul;78(7):e766-e773. doi: 10.4088/JCP.16m11101. PMID 28617566
- [Background] Sinha R, Fox HC, Hong KI, Hansen J, Tuit K, Kreek MJ. Effects of adrenal sensitivity, stress- and cue-induced craving, and anxiety on subsequent alcohol relapse and treatment outcomes. Arch Gen Psychiatry. 2011 Sep;68(9):942-52. doi: 10.1001/archgenpsychiatry.2011.49. Epub 2011 May 2. PMID 21536969
- [Background] Schulte MHJ, Wiers RW, Boendermaker WJ, Goudriaan AE, van den Brink W, van Deursen DS, Friese M, Brede E, Waters AJ. The effect of N-acetylcysteine and working memory training on cocaine use, craving and inhibition in regular cocaine users: correspondence of lab assessments and Ecological Momentary Assessment. Addict Behav. 2018 Apr;79:24-31. doi: 10.1016/j.addbeh.2017.11.044. Epub 2017 Dec 11. PMID 29241082
- [Background] Levi Bolin B, Alcorn JL 3rd, Lile JA, Rush CR, Rayapati AO, Hays LR, Stoops WW. N-Acetylcysteine reduces cocaine-cue attentional bias and differentially alters cocaine self-administration based on dosing order. Drug Alcohol Depend. 2017 Sep 1;178:452-460. doi: 10.1016/j.drugalcdep.2017.05.039. Epub 2017 Jun 29. PMID 28711811
- [Background] Breier A, Liffick E, Hummer TA, Vohs JL, Yang Z, Mehdiyoun NF, Visco AC, Metzler E, Zhang Y, Francis MM. Effects of 12-month, double-blind N-acetyl cysteine on symptoms, cognition and brain morphology in early phase schizophrenia spectrum disorders. Schizophr Res. 2018 Sep;199:395-402. doi: 10.1016/j.schres.2018.03.012. Epub 2018 Mar 24. PMID 29588126
- [Background] Stavro K, Pelletier J, Potvin S. Widespread and sustained cognitive deficits in alcoholism: a meta-analysis. Addict Biol. 2013 Mar;18(2):203-13. doi: 10.1111/j.1369-1600.2011.00418.x. Epub 2012 Jan 20. PMID 22264351

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT04964843/Prot_SAP_ICF_000.pdf